CLINICAL TRIAL: NCT04557072
Title: Selective Versus Nonselective Alpha-blockade Prior to Pheochromocytoma Resection - Systematic Review and Meta-analysis
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Karolina Zawadzka, Principal Investigator, Jagiellonian University
Other Study IDs: SAB vs NAB - pheochromocytoma
Record Dates: First submitted 2020-09-17; First posted 2020-09-21 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Pheochromocytoma
Keywords: pheochromocytoma, surgery, alpha-blockade
MeSH Terms: conditions — Pheochromocytoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The selective alpha-blockade group: Patients treated with selective alpha-blockade before pheochromocytoma surgery
  Interventions: Drug: Selective alpha-1-antagonist
- The non-selective alpha-blockade group: Patients treated with non-selective alpha-blockade before pheochromocytoma surgery
  Interventions: Drug: Non-selective alpha-1-antagonist

INTERVENTIONS:
Drug: Selective alpha-1-antagonist — Patients treated with selective alpha-blockade (prazosin, terazosin, doxazosin)
  Groups: The selective alpha-blockade group
Drug: Non-selective alpha-1-antagonist — Patients treated with non-selective alpha-blockade (phenoxybenzamine)
  Groups: The non-selective alpha-blockade group

SUMMARY:
Our aim was to systematically evaluate the current data on the efficacy of pretreatment with either selective or nonselective alpha-blockade on the hemodynamic instability and morbidity during pheochromocytoma resection.

DETAILED DESCRIPTION:
RCTs and non-randomized controlled studies comparing preoperative selective alpha-blockade (SAB) with nonselective alpha-blockade (NAB) in pheochromocytoma surgery in adults were eligible for inclusion.

All identified articles will be screened by title and abstract. Two independent reviewers will review potentially relevant articles in detail. Dissent will be resolved by consensus and the recommendation of a third observer as required. Data from the included studies will be extracted independently by the two researchers. The Meta-analysis Of Observational Studies in Epidemiology (MOOSE) guidelines will be used for reporting.

Quality of Assessment The Risk Of Bias In Non-randomized Studies - of Interventions (ROBINS-I) tool will be used to assess the quality of included non-randomized studies. The risk of bias of randomized studies will be assessed using the criteria described in the Cochrane Handbook for Systematic Reviews of Interventions .The quality of each study will be assessed by two of the authors. In the event of uncertainties regarding the levels of the studies' quality, a third reviewer will be consulted.

Analysis will be performed using RevMan (Version 5.3, freeware from the Cochrane Collaboration). Odds ratios and their associated 95% confidence intervals will be pooled for dichotomous outcomes using the Mantel-Haenszel random-effects method. Continuous outcomes will be pooled as weighted mean difference (WMD) with 95 per cent confidence interval using the inverse-variance random-effects method. WMD and OR will be presented on the graphs as squares, and pooled WMD and OR will be presented as diamond.

P ≤ 0.05 will be considered a statistically significant difference for hypothesis and P < 0.10 for heterogeneity testing, respectively.

Heterogeneity between the studies will be estimated by statistical tests I2 and Cochran's Q tests.

ELIGIBILITY:
Inclusion Criteria:

* All patients who received selective or nonselective alpha-blockade prior to pheochromocytoma resection

Exclusion Criteria:

* Patients who did not receive alpha blockade
* Patients not undergoing surgery
* No comparison for selective and non-selective pretreatment in the study
* Studies without primary or sufficient data (reviews, guidelines, meeting abstracts, letters),
* Studies reported in a language other than English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RCTs and non-randomized controlled studies comparing preoperative selective α-blockade (SAB) with nonselective α-blockade (NAB) in pheochromocytoma surgery in adults were eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 1344 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Intraoperative maximum systolic blood pressure (mm Hg) | intraoperative

SECONDARY OUTCOMES:
Frequency of systolic blood pressure >160 mmHg | intraoperative
Intraoperative maximum diastolic blood pressure (mm Hg) | intraoperative
intraoperative maximum heart rate (beats/min) | intraoperative
Intraoperative minimum systolic blood pressure (mm Hg) | intraoperative
Intraoperative vasopressors administration | intraoperative
  (number of patients requiring vasopressors administration)
Intraoperative vasodilators administration | intraoperative
  (number of patients requiring vasopressors administration)
Operative time (min) | intraoperative
Overall morbidity | 30 days
Length of hospital stay (days) | Up to 30 days
Postoperative minimum systolic blood pressure (mm Hg) | 24 hours
Postoperative vasopressors administration | 24 hours
  (number of patients requiring vasopressors administration)
Mortality | 30 days
Time of alpha-adrenolytics administration | Up to 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of General Surgery, Jagiellonian University Medical College, Krakow, Polska, Poland